CLINICAL TRIAL: NCT04046003
Title: Tai Chi for Pain Management of Knee Osteoarthritis
Brief Title: Tai Chi for Knee OA Pain Management: a Mechanistic Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Texas Tech University Health Sciences Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Tai Chi for Knee OA pain
Record Dates: First submitted 2019-07-26; First posted 2019-08-06 (Actual); Last update posted 2025-03-28 (Actual); Status verified 2025-03

CONDITIONS: Knee Osteoarthritis; Mind-body Exercise
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Aquatic Therapy

STUDY DESIGN:
Intervention Model Description: 24-form Yang style Tai Chi (60 min/session, 3 sessions/week) for 8 weeks.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Tai Chi intervention (Experimental): 24-form Yang style Tai Chi
  Interventions: Behavioral: Tai chi exercise

INTERVENTIONS:
Behavioral: Tai chi exercise — 24-form Yang style Tai Chi (60 min/session, 3 sessions/week) for 8 weeks

SUMMARY:
This study is to determine how 8-week Tai Chi intervention alters plasma endocannabinoid and its receptors in monocytes/marcrophages, plasma oxylipinds, plasma brain-derived neurotrophic factor, brain white matter connectivity/efficiency, and functional/clinical outcomes in women with knee OA.

DETAILED DESCRIPTION:
Knee osteoarthritis (OA) is one of the five leading causes of disability. Previous studies have shown that a mind-body moderate-intensity Tai Chi (TC) exercise (8-24 weeks) reduced pain and improved physical function for knee OA, when compared to a waiting list, attention control, usual physical activity, or physical therapy. However, TC's mechanisms of action regarding improvement of one's clinical condition and its functional outcomes in individuals with knee OA are poorly understood. This study is to determine how 8-week TC intervention alters plasma endocannabinoid and its receptors in monocytes/marcrophages, plasma oxylipinds, plasma brain-derived neurotrophic factor, brain white matter connectivity/efficiency, and functional/clinical outcomes in women with knee OA.

ELIGIBILITY:
Inclusion Criteria:

1. Postmenopausal women.
2. WOMAC pain score ≥ 50 on at least 1 of the 5 questions in pain subscale (range of 0 to 100, with higher scores indicating greater pain.
3. English literacy.
4. Able to undergo an MRI scan
5. Diagnosed Have the following symptoms associated with knee OA based on American College of Rheumatology clinical classification criteria for osteoarthritis (Peat 2006). Pain in the knee. Need to at least 3 of the following: over 50 years of age, less than 30 minutes of morning stiffness, crepitus on active motion, bony tenderness, bony enlargement, or no palpable warmth of synovium.

Exclusion Criteria:

1. Prior experience with mind-body practice (e.g. TC, Qi Gong, yoga, or acupuncture) or physical therapy programs for knee OA within the past 3 months.
2. Severe medical limitations (i.e., dementia, symptomatic heart or vascular disease, or recent stroke) precluding full participation.
3. Medical/neurologic or other systemic diseases affecting the musculoskeletal systems (i.e. polio/Parkinson's/multiple sclerosis, etc. in addition to cerebral vascular accident or stroke) and diabetes with peripheral neuropathy affecting their sensory/balance.
4. Intra-articular steroid injection or reconstructive surgery on most severely affected knee in the past three months.
5. Intra-articular hyaluronic acid injections on most severely affected knee in the past six months.
6. Inability to walk without an assistive device.

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — Postmenopausal women.
Enrollment: 33 (Actual)
Dates: Start 2019-09-01 (Actual); Primary Completion 2024-06-30 (Actual); Study Completion 2024-08-31 (Actual)

PRIMARY OUTCOMES:
endocannabinoid | Changes from bseline endocannabinoid levels at 8 weeks
  plasma endocannabinoid levels
oxylipins | Changes from baseline oxylipins levels at 8 weeks
  plasma oxylipins levels

SECONDARY OUTCOMES:
endocannabinoid receptors expression | Changes from baseline the affinity of endocannabinoid receptor expression at 8 weeks
  expression of endocannabinoids receptors on peripheral blood mononuclear cells using flow cytometry. Collect venous blood into evacuated tube containing lithium heparin and pour into a Leucosep tube prepared with Ficoll-Paque. Following sequential centrifugation steps, peripheral blood mononuclear cells will be collected and incubate with endotoxin (e.g. LPS or PMA) for 24 hours (Venable 2016). After incubation, PBMC will be collected and stained with cannabinoid receptors (CB1R and CB2R) and markers for monocytes/macrophages (CD14, etc).
BDNF | Changes from baseline BDNF levels at 8 weeks
  plasma brain-derived neurotrophic factor levels using ELISA
white matter connectivity/efficiency of various fiber tracts in the brain | Change from baselinewhite matter connectivity/efficiency of various fiber tracts in the brain at 8 weeks
  We will follow the protocol of Vachon-Presseau et al. 2006 to collect DTI data. DTI images will be acquired using echo planar imaging (72 x 2-mm thick axial slices; matrix size = 128 x 128; ﬁeld of view = 256 x 256mm2, resulting in a voxel size of 2 x 2 x 2mm). Images will have an isotropic distribution along 60 directions using a b-value of 1000s/mm2. For each set of diffusion-weighted data, eight volumes with no diffusion weighting will be acquired at equidistant points throughout the acquisition.
pain sensitivity | Change from baseline pain sensitivity scale at 8 weeks
  We will use quantitative sensory test including windup to assess pain sensitivity in the most painful knee of subject
Pain assessment | Change from baseline pain scale at 8 weeks
  We will use Brief Pain Inventory (questionnaire) for pain assessment.
physical function | Changes from baseline WOMAC results at 8 weeks
  We will use WOAMC questionnaire for physical function assessment
Quality of life assessment | Changes from baseline SF-36 results at 8 weeks
  Quality of life status will be assessed with the Medical Outcomes Study 36-item short form Health Survey (SF-36, version 2), which consists of eight dimensions of health (physical function, bodily pain, general health, vitality, mental health, social function, and role of physical and emotional health) in the conduct of daily activity characteristics will be assessed with self-report SF-36 questionnaires related to self-rated health, depression, anxiety and sleep quality.

CONTACTS AND LOCATIONS:
Overall Officials: Chwan-Li Shen, Principal Investigator — Texas Tech University Health Sciences Center
Locations (1):
- Texas Tech University Health Sciences Center, Lubbock, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Shen CL, Newman JW, Elmassry MM, Borkowski K, Chyu MC, Kahathuduwa C, Neugebauer V, Watkins BA. Tai Chi exercise reduces circulating levels of inflammatory oxylipins in postmenopausal women with knee osteoarthritis: results from a pilot study. Front Med (Lausanne). 2023 Aug 16;10:1210170. doi: 10.3389/fmed.2023.1210170. eCollection 2023. PMID 37654656